CLINICAL TRIAL: NCT03413228
Title: Surveillance of Nosocomial Influenza at Edouard Herriot University Hospital, Lyon, France.
Brief Title: Nosocomial Influenza Surveillance 2018 - 2022
Acronym: NOSOGRIPPE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0868
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Hospital-Acquired Infection; Influenza
MeSH Terms: conditions — Cross Infection; Influenza, Human | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — nasal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Influenza-like illness group
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — An interview to collect some informations will be done: demographic informations, medical history, vaccination against influenza status, symptoms and virological informations. Then, a nasal swab was performed in order to identified the influenza virus.

SUMMARY:
Hospital-acquired influenza is associated with significant morbidity and mortality in hospitalized patients notably elderly patients. Furthermore, it is also associated with a large economic impact for the hospitals.

The transmission of influenza has been mostly reported in pediatric and long-stay units. The chains of transmission of influenza in acute-stay units have to be describe in order to prevent and control potential outbreaks. Furthermore, to know clinical symptoms seems to be important in order to identify potential sources of virus as soon as possible and to set up appropriate hygiene prevention measures. Moreover, the definition of the hospital-acquired influenza has to be harmonized for all over the studies, especially concerning the delay between the admission in the hospital and the symptoms onset.

The aim of this study is to describe the hospital-acquired influenza in a french university hospital of around 800 beds

ELIGIBILITY:
Inclusion Criteria:

* Adult patients and health-care workers in a participating unit in the study,
* more than 18 years old,
* volunteers,
* who present an influenza-like illness defined by fever > 37,8°C or/and cough or sore throat.

Exclusion Criteria:

-Everyone who does not present the inclusion criteria.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Each patient or health-care worker who present ILI (influenza-like illness) at admission or during hospitalization. ILI is defined by fever > 37,8°C or/and cough or sore throat.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients and health-care workers who present an influenza illness. | 5 days maximum
  An interview to collect some informations will be done to evaluate if participants present symptoms of an inflenza illness (fever > 37,8°C or/and cough or sore throat).
  Then, a nasal swab will be performed in order to identified the influenza virus.

CONTACTS AND LOCATIONS:
Locations (1):
- Infection Control unit. Edouard Herriot hospital Lyon - France, Lyon, France

IPD SHARING:
Plan to Share IPD: No